CLINICAL TRIAL: NCT00667641
Title: Phase I Study of Paclitaxel (Taxol) and Bortezomib (Velcade) in Patients With Refractory Solid Tumor Malignancies Involving an Activated MAPK Pathway
Brief Title: Paclitaxel and Bortezomib in Treating Patients With Metastatic or Unresectable Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Vassiliki Karantza-Wadsworth, MD, PhD, UMDNJ/CINJ
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000592905; P30CA072720 (NIH); CINJ-050608; MILLENNIUM-CINJ-050608; CINJ-IRB-0220060270
Record Dates: First submitted 2008-04-25; First posted 2008-04-28 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Breast Cancer; Colorectal Cancer; Head and Neck Cancer; Lung Cancer; Melanoma (Skin); Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent breast cancer; stage IV breast cancer; recurrent prostate cancer; stage IV prostate cancer; recurrent colon cancer; stage IV colon cancer; recurrent pancreatic cancer; stage IV pancreatic cancer; recurrent ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent melanoma; stage IV melanoma; stage IV papillary thyroid cancer; recurrent thyroid cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Melanoma; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Carcinoma, Ovarian Epithelial; Carcinoma, Non-Small-Cell Lung; Thyroid Cancer, Papillary; Thyroid Neoplasms | interventions — Bortezomib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bortezomib — Starting dose level 0.70mg/m2
Drug: paclitaxel — Starting dose level 40mg/m2

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving paclitaxel together with bortezomib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of paclitaxel and bortezomib in treating patients with metastatic or unresectable malignant solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify the maximum tolerated dose of paclitaxel in combination with bortezomib in patients with metastatic or unresectable solid tumor malignancies that involve an activated Ras/Raf/MAPK pathway.

Secondary

* To assess the toxicity of this regimen.
* To assess tumor response in these patients.
* To determine whether Bim is upregulated in peripheral blood mononuclear cells obtained from patients treated with this regimen.
* To correlate markers of Ras/Raf/MAPK pathway activation in fresh or archived tumor tissue with clinical response in these patients.
* To perform pharmacokinetic (PK) studies to determine whether bortezomib alters paclitaxel PK parameters.

OUTLINE: Patients receive paclitaxel IV over 1 hour and bortezomib IV on days 1, 8, and 15. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during course 1 for pharmacokinetic and biomarker studies. Blood samples are analyzed for plasma concentrations of paclitaxel by high performance liquid chromatography and for Bim protein levels and phosphorylation status by western blotting. Tumor tissue samples, if available, are analyzed to evaluate the presence of an activated Ras/Raf/MAPK pathway. Tumor tissue samples are analyzed for Ras and/or Raf mutations by nucleic acid extraction and direct sequencing; Ras and/or Raf overexpression by western blotting; Ras activation assay; and/or phospho-ERK by western blotting and IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor that involves an activated Ras/Raf/MAPK pathway, including the following:

  * Breast cancer
  * Prostate cancer
  * Colon cancer
  * Pancreatic cancer
  * Ovarian cancer
  * Non-small cell lung cancer
  * Melanoma
  * Papillary thyroid cancer
* Metastatic or unresectable disease
* Standard curative or palliative measures do not exist or are no longer effective
* No newly diagnosed, untreated, or uncontrolled brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,500/μL
* WBC ≥ 3,500/μL
* Platelet count ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN (≤ 5 times ULN for tumor involvement of the liver)
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No neuropathy ≥ grade 1 with pain within the past 14 days
* No active infections
* No myocardial infarction within the past 6 months
* No NYHA class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled ventricular arrhythmias
* No evidence of acute ischemia or active conduction system abnormalities by ECG

  * Any ECG abnormality at screening must be documented by the investigator as not medically relevant
* No hypersensitivity to bortezomib, boron, or mannitol
* No serious medical or psychiatric illness likely to interfere with study participation

PRIOR CONCURRENT THERAPY:

* Prior paclitaxel or bortezomib allowed
* At least 4 weeks since prior chemotherapy and/or radiotherapy
* More than 14 days since other prior investigational drugs
* No other concurrent investigational agents
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No concurrent recombinant interleukin-11 (Neumega®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of paclitaxel in combination with bortezomib | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vassil Karantza-Wadsworth, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://www.clinicaltrials.gov/ct2/show/NCT00667641